CLINICAL TRIAL: NCT03145298
Title: A Phase I Study of the Safety and Feasibility of Central Intravenous Delivery of Allogeneic Human Cardiosphere-Derived Stem Cells in Patients With Pulmonary Arterial Hypertension ALPHA Trial
Brief Title: ALlogeneic Cardiosphere-derived Stem Cells (CDCs) for Pulmonary Hypertension therApy
Acronym: ALPHA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Eduardo Marbán, MD, PhD, Director, Cedars-Sinai Heart Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND 16686
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: HPAH (heritable); IPAH (idiopathic); PAH-CTD (connective tissue diseases); PAH-HIV (human immunodeficiency virus)
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Connective Tissue Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study is divided into two portions. The first (Phase 1a) evaluates safety and efficacy of 2 different doses of cells (50 and 100 million cells). The second phase (Phase 1b) takes place after an independent data safety monitoring board has reviewed all the data from Phase 1a and deems it safe and appropriate to proceed to Phase 1b. The latter is a randomized double-blind study in which subjects receive either CAP-1002 or placebo in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Notification of subject randomization will be received by an independent storage/distribution center; the storage/distribution center will have password protected access to the randomization in order to retrieve the treatment assignment. The storage/distribution center will randomly assign an appropriate donor (or placebo) once they receive the designation of active treatment vs. placebo from the interactive system. All Sponsor staff will remain blinded to treatment (CAP-1002 or placebo) assignments. The only time other Sponsor staff will become aware of individual treatments is in the case of an emergency blind break resulting from an SAE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biological: Allogeneic Human Cardiosphere-Derived Cells (CDCs) (Experimental): The Phase 1a portion (N=6 subjects) consists of an open-label, single-arm, study design - dose escalation. The potentially conducted Phase 1b portion of the study (N=20 subjects) consists of a double-blind, randomized, placebo-controlled study design.
  Interventions: Biological: Allogeneic Human Cardiosphere-Derived Stem Cells
- Placebo (Placebo Comparator): The placebo study arm only applies to the Phase Ib portion of the study design. The Phase Ia portion (N=6 subjects) consists of an open-label, single-arm, study design. The potentially conducted Phase Ib portion of the study (N=20 subjects) consists of a double-blind, randomized, placebo-controlled study design with a 1:1 ratio.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Allogeneic Human Cardiosphere-Derived Stem Cells — Human Allogeneic Cardiosphere-Derived Cells is a biologic product consisting largely of cells grown from donated human heart muscle tissue
  Other Names: CAP-1002
  Arms: Biological: Allogeneic Human Cardiosphere-Derived Cells (CDCs)
Biological: Placebo — For use in Phase 1b - Double-blind randomized control portion of the study
  Arms: Placebo

SUMMARY:
Pulmonary Arterial Hypertension or PAH is a progressive condition for which there is no cure. Even with substantial pharmacologic advances in the modern treatment era, survival still remains unacceptably poor, as reported in large PAH registries. Preclinical studies suggest that the administration of allogeneic CDCs have the potential to reduce adverse arteriolar remodeling in PAH which was the basis for the approved investigational new drug (IND). The use of CDCs as an adjunctive therapy in patients comprising 4 sub-groups of patients with PAH in which inflammation and immune dysfunction are key pathophysiologic drivers of PAH.

DETAILED DESCRIPTION:
Patients with IPAH, HPAH, PAH-CTD and PAH-HIV meeting all inclusion and no exclusion criteria will be enrolled. An open label phase 1a study (evaluating dosage and safety) will be conducted. This will followed by a randomized double blind placebo controlled Phase 1b study after Data Safety and Monitoring Board (DSMB) review of the one-month safety data for all the Phase 1a subjects. All patients must have documented PAH diagnosed within the last 5 years and all need to be on stable background PAH specific agents for at least 4 months.

The 4 different etiologies of Pulmonary Arterial Hypertension (PAH) included in this (IND) (IPAH, HPAH, PAH-CTD, PAH-HIV) will be diagnosed based on the following:

i) clinical features and tests to support a diagnosis of PAH: the diagnosis of PAH requires right heart catheterization (RHC) to confirm a hemodynamic profile compatible with PAH. This includes a mean pulmonary artery pressure (PAP) ≥ than 25 mmHg at rest, with a pulmonary capillary wedge pressure < 15 mmHg. (If slightly elevated, will confirm with LVEDP measure as is our usual standard of care) and pulmonary vascular resistance (PVR) of > 3 Wood units. In addition, there should be no features to suggest other associations for PAH (also included in Group 1) or evidence to suggest PAH owing to left heart disease (Group 2), PH due to lung diseases (Group 3), Chronic thromboembolic pulmonary hypertension (Group 4) or miscellaneous disorders of unclear mechanism ii) clinical features and tests to support a specific designation of each subset of PAH:

* Idiopathic PAH (IPAH): This is a diagnosis of exclusion in which a firm diagnosis of PAH is made and there are no other etiologies or associations determined that fall into Group 1
* Heritable PAH (HPAH): This diagnosis is based on a family history of PAH with or without a documented genetic mutation associated with PAH (such as BMPR2 mutations that are present in up to 75% of HPAH patients). No other PAH association is present.
* PAH - Connective Tissue Disease (PAH-CTD): These patients have a confirmed diagnosis of PAH as well as firm evidence to support a diagnosis of a connective tissue disease. In the REVEAL registry, scleroderma-associated PAH accounted for 60% of PAH-CTD . All PAH-CTD cases will be referred by or evaluated by a rheumatologist to ensure a firm diagnosis. While all CTDs can be complicated by PAH, the most common associations are described below.

  1. Scleroderma (SSc): We use the ACR/EULAR criteria for the diagnosis and classification of systemic sclerosis. Patients with SSc-APAH may exhibit features of limited scleroderma, such as, calcinosis, Reynaud's, esophageal dysmotility, sclerodactyly (with skin thickening of the fingers of both hands extending proximal to the metacarpophalangeal joints) and telangiectasia. In those with limited scleroderma anticentromere antibodies are commonly positive. In patients with diffuse cutaneous scleroderma, SSc-PAH can also be seen. They exhibit diffuse skin thickening and tightening. Anti-topoisomerase antibodies (anti Scl70) may be positive but interestingly, their absence is more likely to be associated with PAH. Other autoantibodies that are associated with an increased risk of SSc-PAH include anti-U1-ribonucleoprotein antibodies (RNP), nucleolar pattern of anti-nuclear antibody (nucleolar-ANA), and rarely antiphospholipid antibodies.
  2. Systemic Lupus Erythematosus (SLE): We use the Systemic Lupus International Collaborating Clinics (SLICC) classification, which requires at least 4/17 criteria including at least 1 clinical criterion and 1 immunologic criterion or biopsy proven lupus nephritis. On history and physical exam, the following are highly suggestive: Photosensitive skin lesions (malar rash or discoid lesions), painless ulcers (oral or nasal), features of a serositis, alopecia, Raynaud's, arthralgia/arthritis (often migratory) etc. Immunologic antibody studies included in SLICC are: Positive ANA, anti-dsDNA, anti-Sm, antiphospholipid, low complement, positive direct Coombs test.
  3. Mixed Connective Tissue Disease (MCTD): This is characterized by overlapping features of SLE, SSc and polymyositis (PM), as well as high titers of anti-U1 ribonucleoprotein (RNP). The old term for this is anti-extractable nuclear protein (anti-ENA).
  4. Rheumatoid Arthritis (RA): RA is a symmetrical distal inflammatory poly arthritis condition. The criteria developed and validated by the American College of Rheumatology (ACR) has been used in numerous drug studies which requires at least four of these seven criteria for diagnosis (morning stiffness, arthritis of three or more joint areas, arthritis of the hands, symmetric arthritis, rheumatoid nodules and classic radiographic erosive changes). Immunologic studies include positive rheumatoid factor (RF) and anti-cyclic citrullinated peptide (CCP) antibody.
* PAH- Human Immunodeficiency Virus (HIV): Patients will have a firm diagnosis with positive HIV testing (i.e. positive 4th generation immunoassay and positive confirmatory testing such as Western Blot or HIV-1/HIV-2 antibody differentiation immunoassay) and managed by an infectious disease/HIV specialist. These patients have hemodynamic criteria for PAH present, but the only association on workup is the presence of HIV.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of IPAH, HPAH, PAH-CTD, PAH-HIV
* NYHA Functional Class: II or III
* 6MWD > 150 m
* Able to maintain O2 saturation at rest ≥ 90% (with or without supplemental O2). O2 use during the course of the study is permitted.
* The subjects must be on PAH-specific therapies for at least 4 months and on a stable dose for at least 4 weeks prior to enrollment into study. PAH-specific agents can include: prostanoids, prostacyclin receptor agonist, endothelin receptor antagonists, phosphodiesterase-5 inhibitors and soluble guanylate cyclase stimulator agents alone or in combination
* All patients with PAH-HIV must be on a stable and effective HAART combination regimen
* Pulmonary capillary wedge pressure (PCWP) or LVEDP < 15 mm Hg
* Age: 18 -75 years
* Ability to provide informed consent and follow-up with protocol procedures

Exclusion Criteria:

* Diagnosis of PAH other than IPAH, HPAH, PAH-CTD or PAH-HIV
* Right atrial pressure > 20 mmHg as measured by right heart catheterization (RHC) on day of pre-infusion
* History of clinically-significant coronary artery disease, including myocardial infarction, coronary stent placement or coronary artery bypass surgery within the previous 5 years, LV dysfunction
* History or demonstration of significant ventricular tachy-arrhythmias or conduction abnormalities
* Significant interstitial lung disease (on imaging and PFTs; FVC: < 60%;
* Chronic thromboembolic pulmonary hypertension (CTEPH)
* Estimated glomerular filtration rate (GFR) ≤ 50 mL/min
* Active uncontrolled infection
* Non-pulmonary vascular disease with life expectancy of < 3 years
* Hypersensitivity to contrast agents
* Active allergic reactions
* History of previous stem cell therapy
* Participation in an on-going protocol studying an experimental drug or device
* Current alcohol or drug abuse because of anticipated difficulty in complying with protocol-related procedures
* Pregnant/nursing women as well as men and women of child-bearing potential without use of active and highly reliable contraception
* Known history of viral hepatitis
* Abnormal liver function (transaminases > 3 times the upper reference range; total bilirubin > 2 times the upper reference range without a reversible, identifiable cause
* Evidence of tumor on screening of chest/abdominal/pelvic (body) CT scan
* History of malignancy within the last 5 years, except for resected skin basal cell or squamous cell carcinoma, treated cervical dysplasia or treated in-situ cervical cancer grade 1
* Any prior organ transplant
* Being actively listed for, or under active consideration for, an organ transplant of any kind, including lung transplantation
* Known hypersensitivity to bovine products
* Known hypersensitivity to dimethyl sulfoxide (DMSO)
* Any condition or treatment which (in the opinion of investigator), places the patient at an unacceptable risk if enrolled
* Patients with PAH-HIV will be excluded with any of the following clinical conditions:

  * CD4 T-cell count < 200 /mm3 within 90 days prior to screening
  * A detectable viral load within 90 days prior to screening
  * Active opportunistic infections within 90 days prior to screening
  * Changes in antiretroviral regimen within 90 days prior to screening
* Significant anemia or a falling Hb would make patient ineligible. Platelet counts ≤ 100,000/mm3 and absolute neutrophil count < 1,500/mm3 excludes the patient
* History of heparin induced thrombocytopenia (HIT) (unless current HIT Panel is negative)

NOTE: Those eligible individuals who have had four or more previous gadolinium contrast scans will have a cardiac MRI without contrast

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Primary Safety (Early) endpoints including the determination of Gas Exchange and Hemodynamics; Detection of Arrhythmias; Sudden unexpected death and Mortality and Morbidity | Within 72 hours of infusion
  * Determination of Gas Exchange: Significant hypoxemia within the 1st 72 hours following the infusion of CAP-1002 cells as determined by arterial blood gas analysis or pulse oximetry on or off O2, which is a distinct change from values obtained at screening. (PaO2 < 55mmHg; SPO2 < 85%).
  * Determination of Hemodynamics: Significant tachycardia and hypotension; while PA cath in-situ: fall in cardiac output; significant rise in PA systolic pressure, mean right atrial pressure. Note, hemodynamic measurements will be obtained, as clinically indicated over a 1-hour time frame post CDC infusion. If the patient is deemed stable after this 1-hour time frame, the PA catheter will be withdrawn in the cardiac catheterization laboratory, and the patient will be transferred to the ICU for further monitoring.
  * Detection of Arrhythmias: development of supra-ventricular tachyarrhythmias

SECONDARY OUTCOMES:
Secondary Safety (Long Term) endpoints including ongoing monitoring of events listed for primary safety endpoints as well as long term monitoring for a composite of time to clinical worsening. | One year
  Clinical Worsening is described as:
  * Death (all-cause mortality)
  * Hospitalization for worsening PAH:
  * Non-elective hospitalization for ≥ 24 hours
  * Signs and symptoms of RV failure to include one or more of: increased dyspnea, clinically significant deterioration in exercise capacity, syncope or pre-syncope, hypoxemia, edema, hepatomegaly, ascites
  * Initiation of parenteral prostanoids or chronic O2 therapy if not previously receiving
  * Decrease in Functional Class:
  * ≥ 15% reduction in 6MWD from screening (confirmed on 2 tests on different
  * days over 2 weeks)
  * Need for additional PAH-specific therapy
  * Progressive disease requiring balloon atrial septostomy +/- lung transplantation
Exploratory Secondary Efficacy Endpoints measuring right ventricular function and pressure estimates | One year
  Transthoracic Echo (TTE):
  * Tricuspid annular plane systolic excursion (TAPSE)
  * RV (Right Ventricular) Fractional Area Change
  * Tricuspid Tissue Doppler Velocity
  * Pulmonary and right atrial pressure estimates
  Right Heart Catheterization:
  * Right atrial pressure (RAP)
  * RV systolic, diastolic pressures
  * PA systolic, diastolic and mean pressures
  * Pulmonary capillary wedge pressure
  * Total pulmonary arterial compliance
  * Cardiac Output (CO)/Cardiac Input (CI)

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Lewis, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Uncertain